CLINICAL TRIAL: NCT02805634
Title: Correlation Between the 'Nine Holes Peg Test' Performance and the Triple Stimulation Technique Within a Group a Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Bernard Dachy, Head of clinic, Brugmann University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-TST02
Record Dates: First submitted 2016-03-31; First posted 2016-06-20 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
Keywords: nine holes peg; triple stimulation; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple sclerosis (Experimental): Patients with multiple sclerosis, followed by Dr Dachy within the CHU Brugmann Hospital.
  Interventions: Other: Nine Hole Test; Device: Triple Stimulation Technique
- Control group (Other): Control group without neurological pathology
  Interventions: Other: Nine Hole Test; Device: Triple Stimulation Technique

INTERVENTIONS:
Other: Nine Hole Test — The Nine Hole Pegs technique is a simple manual dexterity test, commonly used in ergotherapy. The participant tries to place 9 pegs in a 9 holes perforated plate, and then tries to remove them as quickly as possible. The hand must stay in a depression within the plate, thereby insuring a constant distance between the hand and the pegs.
Device: Triple Stimulation Technique — TST (Triple stimulation technique) combines two techniques used in neurologic diagnosis: magnetic stimulation and electroneuromyography. It is based on the principle of two collisions between the descending central stimulation (magnetic stimulation) and the ascending peripheric stimulation. TST allows to better quantify central nervous system diseases. The abnormal amplitude registered by TST is proportional to the intensity of conduction disorders. The evaluation of these disorders is more precise than with the magnetic stimulation technique alone.

SUMMARY:
The main goal of this study is to determine if the Triple Stimulation Technique (TST) can be correlated to performance in the manual dexterity 'nine holes peg' test, within a control group and a group of patients with multiple sclerosis.

TST (Triple stimulation technique) combines two techniques used in neurologic diagnosis: magnetic stimulation and electroneuromyography. It is based on the principle of two collisions between the descending central stimulation (magnetic stimulation) and the ascending peripheric stimulation. TST allows to better quantify central nervous system diseases. The abnormal amplitude registered by TST is proportional to the intensity of conduction disorders. The evaluation of these disorders is more precise than with the magnetic stimulation technique alone.

The Nine Hole Pegs technique is a simple manual dexterity test, commonly used in ergotherapy. The participant tries to place 9 pegs in a 9 holes perforated plate, and then tries to remove them as quickly as possible. The hand must stay in a depression within the plate, thereby insuring a constant distance between the hand and the pegs.

The nine hole peg will be realized first, and the triple stimulation examination performed after. The acquired data will be analyzed in order to find a correlation between the impairment level given by these two tests.

ELIGIBILITY:
Inclusion Criteria:

Control group:

* No history of neurological disease
* No medicines intake that could disturb performance within the tests (psychotropic medications, sedatives, anti spastic and drugs acting on neuromuscular transmission).

Multiple sclerosis group

* Multiple sclerosis diagnose. Patients followed by Dr Dachy, within the CHU Brugmann Hospital.

Exclusion Criteria:

* Persons carrying ferromagnetic material (implants, pacemaker).
* Epilepsy history.
* Patients who have had a head trauma with loss of consciousness and/or brain injury.
* Pregnant woman.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Amplitude of the motor evoked potentials | during the TST (30 min)
Amplitude ratio of the TST | during the TST (30 min)
Surface ratio of the TST | during the TST (30 min)
Nine Holes Peg test result | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Bernard, MD, Principal Investigator — CHU Brugmann; Pedro Calderon, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Magistris MR, Rosler KM, Truffert A, Myers JP. Transcranial stimulation excites virtually all motor neurons supplying the target muscle. A demonstration and a method improving the study of motor evoked potentials. Brain. 1998 Mar;121 ( Pt 3):437-50. doi: 10.1093/brain/121.3.437. PMID 9549520
- [Background] Magistris MR, Rosler KM, Truffert A, Landis T, Hess CW. A clinical study of motor evoked potentials using a triple stimulation technique. Brain. 1999 Feb;122 ( Pt 2):265-79. doi: 10.1093/brain/122.2.265. PMID 10071055
- [Background] Buhler R, Magistris MR, Truffert A, Hess CW, Rosler KM. The triple stimulation technique to study central motor conduction to the lower limbs. Clin Neurophysiol. 2001 May;112(5):938-49. doi: 10.1016/s1388-2457(01)00506-5. PMID 11336912
- [Background] Humm AM, Beer S, Kool J, Magistris MR, Kesselring J, Rosler KM. Quantification of Uhthoff's phenomenon in multiple sclerosis: a magnetic stimulation study. Clin Neurophysiol. 2004 Nov;115(11):2493-501. doi: 10.1016/j.clinph.2004.06.010. PMID 15465437
- [Background] Humm AM, Z'Graggen WJ, von Hornstein NE, Magistris MR, Rosler KM. Assessment of central motor conduction to intrinsic hand muscles using the triple stimulation technique: normal values and repeatability. Clin Neurophysiol. 2004 Nov;115(11):2558-66. doi: 10.1016/j.clinph.2004.06.009. PMID 15465445
- [Background] Humm AM, Z'Graggen WJ, Buhler R, Magistris MR, Rosler KM. Quantification of central motor conduction deficits in multiple sclerosis patients before and after treatment of acute exacerbation by methylprednisolone. J Neurol Neurosurg Psychiatry. 2006 Mar;77(3):345-50. doi: 10.1136/jnnp.2005.065284. Epub 2005 Sep 20. PMID 16174651
- [Background] Rosler KM, Scheidegger O, Magistris MR. Corticospinal output and loss of force during motor fatigue. Exp Brain Res. 2009 Aug;197(2):111-23. doi: 10.1007/s00221-009-1897-z. Epub 2009 Jul 2. PMID 19572125
- [Background] Andersen B, Westlund B, Krarup C. Failure of activation of spinal motoneurones after muscle fatigue in healthy subjects studied by transcranial magnetic stimulation. J Physiol. 2003 Aug 15;551(Pt 1):345-56. doi: 10.1113/jphysiol.2003.043562. Epub 2003 Jun 24. PMID 12824449
- [Background] Attarian S, Verschueren A, Pouget J. Magnetic stimulation including the triple-stimulation technique in amyotrophic lateral sclerosis. Muscle Nerve. 2007 Jul;36(1):55-61. doi: 10.1002/mus.20789. PMID 17443663
- [Background] Tan F, Wang X, Li HQ, Lu L, Li M, Li JH, Fang M, Meng D, Zheng GQ. A randomized controlled pilot study of the triple stimulation technique in the assessment of electroacupuncture for motor function recovery in patients with acute ischemic stroke. Evid Based Complement Alternat Med. 2013;2013:431986. doi: 10.1155/2013/431986. Epub 2013 Jun 10. PMID 23840255
- [Background] Oxford Grice K, Vogel KA, Le V, Mitchell A, Muniz S, Vollmer MA. Adult norms for a commercially available Nine Hole Peg Test for finger dexterity. Am J Occup Ther. 2003 Sep-Oct;57(5):570-3. doi: 10.5014/ajot.57.5.570. PMID 14527120
- [Background] Chan T. An investigation of finger and manual dexterity. Percept Mot Skills. 2000 Apr;90(2):537-42. doi: 10.2466/pms.2000.90.2.537. PMID 10833751
- [Background] Kellor M, Frost J, Silberberg N, Iversen I, Cummings R. Hand strength and dexterity. Am J Occup Ther. 1971 Mar;25(2):77-83. No abstract available. PMID 5551515
- [Background] Chen HM, Chen CC, Hsueh IP, Huang SL, Hsieh CL. Test-retest reproducibility and smallest real difference of 5 hand function tests in patients with stroke. Neurorehabil Neural Repair. 2009 Jun;23(5):435-40. doi: 10.1177/1545968308331146. Epub 2009 Mar 4. PMID 19261767
- [Background] Earhart GM, Cavanaugh JT, Ellis T, Ford MP, Foreman KB, Dibble L. The 9-hole PEG test of upper extremity function: average values, test-retest reliability, and factors contributing to performance in people with Parkinson disease. J Neurol Phys Ther. 2011 Dec;35(4):157-63. doi: 10.1097/NPT.0b013e318235da08. PMID 22020457
- [Background] Erasmus LP, Sarno S, Albrecht H, Schwecht M, Pollmann W, Konig N. Measurement of ataxic symptoms with a graphic tablet: standard values in controls and validity in Multiple Sclerosis patients. J Neurosci Methods. 2001 Jul 15;108(1):25-37. doi: 10.1016/s0165-0270(01)00373-9. PMID 11459615